CLINICAL TRIAL: NCT02985242
Title: SGLT2-inhibition With Empagliflozin Reduces Progression of Diabetic Retinopathy in Patients With High Risk of Diabetic Macular Edema (The SUPER-Trial)
Brief Title: Empagliflozin Reduces Progression of Diabetic Retinopathy in Patients With High Risk of Diabetic Macular Edema
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulties to recruit planned numbers of patients within reasonable time frame
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-04EMPA-EYE; 2016-000825-38 (EudraCT Number)
Record Dates: First submitted 2016-11-25; First posted 2016-12-07 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin/glimepiride placebo (Experimental): Empagliflozin 25 mg film-coated tablet p.o. daily and glimepiride matching placebo p.o. daily
  Duration of treatment: 12 months
  Interventions: Drug: Empagliflozin; Drug: Glimepiride placebo
- Glimepiride/empagliflozin placebo (Active Comparator): Glimepiride 2 mg tablet p.o. daily and empagliflozin matching placebo p.o. daily
  Duration of treatment: 12 months
  Interventions: Drug: Glimepiride; Drug: Empagliflozin placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin film-coated tablet
  Arms: Empagliflozin/glimepiride placebo
Drug: Glimepiride — Glimepiride tablet
  Arms: Glimepiride/empagliflozin placebo
Drug: Empagliflozin placebo — Placebo tablet manufactured to mimic Empagliflozin 25 mg film-coated tablet
  Arms: Glimepiride/empagliflozin placebo
Drug: Glimepiride placebo — Placebo tablet manufactured to mimic Glimepiride 2 mg tablet
  Arms: Empagliflozin/glimepiride placebo

SUMMARY:
This is a prospective, randomized, active control, two-arm parallel, double-blind, monocenter phase IV clinical trial. The trial compares empagliflozin to glimepiride in patients with type 2 diabetes mellitus in addition to standard of care treatment.

Patients with type 2 diabetes mellitus who are between 18 and 80 years of age will be recruited for the clinical trial and randomly allocated to either receive empagliflozin or glimepiride.

The assumption of the study is that empagliflozin slows down diabetic retinopathy progression rate and thus a lower microaneurysm formation rate compared to subjects treated with glimepiride by substantially decreased cellular glucotoxicity will be achieved.

ELIGIBILITY:
Inclusion Criteria:

1. women and men between 18 - 80 years of age
2. type 2 diabetes mellitus
3. early to moderate stage diabetic retinopathy (ETDRS: 20 (microaneurysms only) to 35 (microaneurysms/ hemorrhages and/or hard exsudates)) in one or both eyes
4. stable HbA1c (± 0.5%) for at least 12 weeks
5. antidiabetic treatment with either diet, metformin, DPP4, GLP1, pioglitazone, acarbose, or respective combinations
6. HbA1c ≥ 6.5 and ≤ 10.0 %
7. body mass index < 46 kg/m2
8. office blood pressure ≤ 150/95 mmHg (confirmed on a second day; 24h ambulatory blood pressure measurement (ABPM) is allowed to check accuracy of office values; inclusion with 24h mean blood pressure ≤ 145/90 mm Hg is possible); patients with hypertension should be treated according to current treatment guidelines
9. either women without childbearing potential defined by:

   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy
   * hysterectomy
   * ≥ 50 years and in postmenopausal state > 1 year
   * < 50 years and in postmenopausal state > 1 year with serum follicle stimulating hormone (FSH) > 40 IU/l and serum estrogen < 30 ng/l or a negative estrogen test, both at screening or women of childbearing potential with a negative serum beta human chorionic gonadotropin (ß-hCG) pregnancy test at screening who agree to meet one of the following criteria from the time of screening, during the study and for a period of 4 days following the last administration of study medication:
   * correct use of one of the following accepted contraception methods: hormonal contraceptives (combined oral contraceptives, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), intrauterine device (IUD/IUS) or a double barrier method, e.g. condom and occlusive cap (diaphragm or cervical/vault caps) with spermicide (foam, gel, film, cream or suppository)
   * true abstinence (periodic abstinence and withdrawal are not acceptable methods of contraception)
   * sexual relationship only with female partners
   * sterile male partners
10. signed written informed consent and willingness to comply with treatment and follow-up procedures
11. capability of understanding the investigational nature, potential risks and benefits of the clinical trial

Exclusion Criteria:

1. Type 1 diabetes
2. uncontrolled diabetes mellitus type 2 with fasting glucose > 13.3 mmol/l confirmed on a second day
3. known or suspected hypersensitivity to empagliflozin, glimepiride, or any excipients; and / or known or suspected hypersensitivity to sulfonylureas, sulfonamides or SGLT2 inhibitors in general
4. history of multiple severe hypoglycemic episodes within the last two years
5. use of Insulin, SGLT2-inhibitor, sulfonylurea derivate or a glinide within past 3 months
6. clinical significant macular edema in both eyes and indication for intravitreal anti-VEGF treatment for both eyes at screening or baseline visit. Eyes with a small amount of intraretinal or subretinal fluid (seen in OCT) but no need for intravitreal treatment as judged by the investigator (according to current practice patterns) may be included. Eyes with a history of intravitreal treatment of macular edema which do not need ongoing intravitreal treatment at the time of screening may be included.
7. eye diseases or pathologies that prevent clear ophthalmoscopy and evaluation of study parameters, thus not allowing study participation according to the investigator´s judgment, such as (but not only) vitreous hemorrhage, mature cataract, macular pathologies other than diabetic maculopathy
8. history of ketoacidosis or metabolic acidosis
9. use of loop diuretics
10. history of > 1 urogenital infection/year
11. any history of stroke, transient ischemic attack (TIA), instable angina pectoris or myocardial infarction within last 3 months prior to baseline visit
12. congestive heart failure New York Heart Association (NYHA) III and IV
13. severe valvular or left ventricular outflow obstruction disease needing intervention;
14. atrial fibrillation/flutter with a mean ventricular response rate at rest >100 beats per minute
15. chronic lower urinary tract infections (but not simple asymptomatic bacteriuria)
16. eGFR < 60 ml/min/1,73 m2 (MDRD-formula, confirmed on a second day)
17. chronic diarrhea, any clinical signs of volume depletion or a hematocrit > 48 % (women) and > 53 % (men)
18. elevated risk for volume depletion, e.g. history of severe volume depletion that required medical therapy
19. chronic liver disease (including known active hepatitis) and/or screening alanine transaminase (ALT) or aspartate transaminase (AST) > 3 x upper limit of normal (ULN) (confirmed on a second day)
20. Subjects with known seropositivity to human immunodeficiency virus.
21. acute illness at screening or randomization according to judgement by the investigator or patient
22. drug or alcohol abuse
23. psychosomatic or psychiatric diseases requiring hospitalization during the last 12 months
24. clinical evidence of current malignancy with exception of basal cell or squamous cell carcinoma of the skin, and cervical intraepithelial neoplasia (5 years prior to randomization)
25. any medical or surgical intervention planned for the next 13 months after randomization not allowing study participation according to the investigator´s judgment
26. current participation in any other clinical trial or participation in another clinical trial within 30 days before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Microaneurysm formation rate over 12 months, i.e. number of newly developed microaneurysms within 12 months | Weeks 27 and 52

SECONDARY OUTCOMES:
Change in diabetic retinopathy stage (≥ 2 step change on ETDRS severity score) | Weeks 27 and 52
Change in microaneurysm count | Weeks 27 and 52
Microaneurysm formation rate after 6 months (compared to baseline) | after 6 months
Change in retinal thickness (as measured by Optical Coherence Tomography) | Weeks 27 and 52
Change in retinal perfusion of microvasculature within the retina (flow in Optical Coherence Tomography Angiography) | Weeks 27 and 52
Progression to clinically significant macular edema (CSME) | Up to 52 weeks
Change in intraocular lipid content (hard exsudates) | Weeks 27 and 52
Change in composite clinical outcome evaluating progression to proliferative diabetic retinopathy (PDR) based on photography, angiography plus clinically important events defining PDR (e.g. vitreous haemorrhage) | Weeks 27 and 52
Change in best corrected visual acuity (BCVA [ETDRS letters]) | Weeks 27 and 52
Change in HbA1c | Weeks 2, 7, 12, 17, 22, 27, 32, 37, 42, 47, 52 and 55
Change in fasting glucose | Weeks 2, 7, 12, 17, 22, 27, 32, 37, 42, 47, 52 and 55
Change in body weight and body fat mass | Weeks 27, 52 and 55
Change in ambulatory blood pressure | Weeks 27 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Pielen, MD, Principal Investigator — Hannover Medical School, University Eye Hospital
Locations (1):
- Hannover Medical School, University Eye Hospital and CRC Core Facility Hannover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No